CLINICAL TRIAL: NCT00179712
Title: Phase I/II Open-Label, Dose Escalation Study To Determine The Maximum Tolerated Dose And To Evaluate The Safety Profile of Lenalidomide (Revlimid®) With Topotecan In Subjects With Advanced Ovarian and Primary Peritoneal Carcinoma
Brief Title: Study of Lenalidomide With Topotecan In Subjects With Advanced Ovarian and Primary Peritoneal Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Prologue Research International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: CC-5013-OVRY-002
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Ovarian Cancer
Keywords: cc-5013; revlimid; ovarian cancer; celgene
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Lenalidomide; Topotecan

INTERVENTIONS:
Drug: CC-5013
Drug: topotecan

SUMMARY:
Phase I will determine the MTD and evaluated the safety profile of oral lenalidomide on days 1-14 when given with topotecan on days 1-5 of every 21 day cycle Phase II will commence once the MTD is established, additional subjects will be enrolled and receive oral lenalidomide on days 1-14 with topotecan on days 1-5 in 21 day cycles until disease progression is documented.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must understand and voluntarily sign an informed consent document.
2. Age >or = to 18 years at the time of signing informed consent form.
3. Subjects must be able to adhere to the study visit schedule and other protocol requirements.
4. Histological or cytological documentation of advanced ovarian or primary peritoneal carcinoma.
5. Radiographic or clinical evidence of measurable metastatic advanced ovarian or primary peritoneal carcinoma. Subjects must have measurable disease at least 2 cm in diameter.
6. Subjects must have been treated and progressed following chemotherapy which includes platinum and paclitaxel.
7. ECOG performance status of 0 or 1 (Appendix I: ECOG Performance Status Scale).

Exclusion Criteria:

1. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1,500 cells/mm3 (1.5 x 109/L)
   2. Platelet count <100,000 cells/mm3 (100 x 109/L)
   3. Serum creatinine >1.5 mg/dL (133 mmol/L)
   4. Serum SGOT/AST or SGPT/ALT >3.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >2.0 mg/dL (34 mmol/L)
2. Any serious medical condition or psychiatric illness that places the subject at an unacceptable risk for study participation or would prevent the subject from signing the informed consent.
3. Prior history of malignancy (except basal cell or squamous cell carcinoma or carcinoma in situ of the breast) unless the subject has been free of disease for > 1 year.
4. Known brain or leptomeningeal disease (CT scan or MRI of the brain required only in case of clinical suspicion of central nervous system involvement).
5. More than 1 prior chemotherapy regimen. However, subjects with platinum sensitive disease (i.e., subjects who fail a platinum containing regimen at least six months after completing the regimen) who are retreated with a platinum containing regimen are eligible.
6. Concurrent use of any other anti-cancer agents.
7. Any prior use of lenalidomide.
8. Prior > or = to grade 3 (see Appendix III) rash or any desquamating (blistering) rash while taking thalidomide.
9. Prior . Or = to grade 3 (see Appendix III) allergic reaction/hypersensitivity to thalidomide.
10. Use of any standard or experimental anti-cancer drug therapy within 28 days of the initiation of study drug therapy.
11. Known active Hepatitis C.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-04; Study Completion 2006-11

PRIMARY OUTCOMES:
Phase I-To determine the MTD and evaluate the safety profile of oral lenalidomide and topotecan
Phase II-To explore the anti-tumor activity based on objective response rate (CR + PR) of the combination of oral lenalidomide and topotecan

SECONDARY OUTCOMES:
Phase I-To explore the anti-tumor activity based on response of the combination of lenalidomide and topotecan.
Phase II-To explore the safety profile of the combination of lenalidomide and topotecan

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medical College of GeorgiaDept of OBGYN, Augusta, Georgia
  - University of MinnesotaObstetrics & Gynecology, MMC, Minneapolis, Minnesota
  - Ohio State University, Columbus, Ohio

REFERENCES:
- [Background] Carter JS, Downs LS Jr. A prospective clinical trial of lenalidomide with topotecan in women with advanced epithelial ovarian carcinoma. Int J Clin Oncol. 2011 Dec;16(6):666-70. doi: 10.1007/s10147-011-0243-1. Epub 2011 May 10. PMID 21556801